CLINICAL TRIAL: NCT00117299
Title: A Phase II, Open-Label Study of PTK787/ZK222584 in the Treatment of Metastatic Gastrointestinal Stromal Tumors (GISTs) Resistant to Imatinib Mesylate
Brief Title: PTK787/ZK222584 in the Treatment of Metastatic Gastrointestinal Stromal Tumors Resistant to Imatinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Bayer (Industry)
Responsible Party: Heikki Joensuu, Helsinki University central Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPTK787 A2401/300267; GIST PTK787/ZK222584
Record Dates: First submitted 2005-06-30; First posted 2005-07-06 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Sarcoma
Keywords: Gastrointestinal stromal tumor; GIST; Sarcoma; PTK787; ZK 222584; Tyrosine kinase inhibitor; Tyrosine kinase; VEGF; Vascular endothelial growth factor; VEGFR; Vascular endothelial growth factor receptor; KDR; KIT; c-KIT; Platelet derived growth factor receptor; PDGFR
MeSH Terms: conditions — Sarcoma; Gastrointestinal Stromal Tumors | interventions — vatalanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): PTK/ZK o.d. 1250 mg p.o.
  Interventions: Drug: PTK787/ZK222584

INTERVENTIONS:
Drug: PTK787/ZK222584 — PTK787/ZK222584 is administered at the dosage of 1250 mg o.d. orally
  Other Names: vatalanib

SUMMARY:
This study evaluates the safety and efficacy of a novel tyrosine kinase inhibitor, PTK787/ZK222584, in the treatment of GIST (gastrointestinal stromal tumor) that is resistant to imatinib mesylate (Gleevec). The study participants are required to have histologically confirmed GIST with prior imatinib treatment for metastatic GIST. is administered orally 1250 mg/day. Six patients will first enter the study. If clinical benefit is obtained in >1 of 6 patients, 9 and 30 additional patients will be entered into the protocol in two stages (a maximum of 45 patients will be entered). Patients who benefit from the study treatment will be treated with PTK787/ZK222584 until treatment failure.

DETAILED DESCRIPTION:
This is an open-label, phase II study of PTK787/ZK222584 designed to determine the safety and efficacy of PTK787/ZK222584 in the treatment of imatinib-resistant GIST. The PTK787/ZK222584 dose used is 1250 mg daily. Six patients will first enter the study using a two-stage approach. If clinical benefit is obtained in >1 of 6 patients, 9 and 30 additional patients will be entered into the protocol (a maximum total number of 45 patients will be entered). Clinical benefit is defined as the occurrence of one or more of the following 3 measures: 1) objective response to PTK787 (a confirmed or unconfirmed partial response [PR] or a complete response [CR]); 2) metabolic response defined as >50% decrease in the standardized uptake value (SUV) of FDG uptake in >1 FDG-avid lesions in one or more of the patients; or 3) stabilized disease for 3 months or longer accompanied by symptomatic or performance status improvement. Medical history, current medical conditions, weight, height, and an electrocardiogram are recorded prior to the study entry. Other baseline examinations include a chest X-ray, hematologic tests, a coagulation panel, serum chemistries, urine analysis, a serum pregnancy test and a radiological assessment of the tumor. Tumor response is monitored with imaging at 4- to 8-week intervals. Hematological tests and serum chemistries are evaluated at 1- to 4-week intervals, and adverse events are collected continuously. Research blood tests are collected at the times of tumor evaluations. Dose adjustments are carried out as per the protocol. Patients who benefit from the study treatment will be treated with PTK787/ZK222584 until treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed GIST
* Imatinib resistance (primary resistance with progression, or progression after initial response). Resistance is defined as objective evidence of progression after at least 4 weeks of treatment with imatinib.
* Imatinib therapy has been interrupted >7 days before study entry
* Metastatic disease confirmed histologically, cytologically or radiologically
* Presence of measurable tumor lesions as determined by RECIST criteria
* Age 18 years or older
* WHO performance status of 2 or less
* Blood neutrophil count (ANC) 1.5 x 10^9/L or higher
* Platelet count 100 x 10^9/L or higher
* Serum bilirubin 1.5 x ULN (upper limit of normal) or less
* Serum creatinine 2.0 x ULN or less
* Written informed consent obtained according to local guidelines

Exclusion Criteria:

* Patients who have received chemotherapy less than 4 weeks prior to entry into this study or who have not recovered from side effects of such therapy
* Patients who have received a cumulative dose of doxorubicin >450 mg/m2 or epirubicin 800 mg/m2
* Patients who have received immunotherapy within 2 weeks or who have not recovered from side effects of such therapy
* Patients who have received radiotherapy within 2 weeks or who have not recovered from side effects of such therapy
* Major surgery within 2 weeks prior to entry into this study or patients who have not recovered from side effects of such therapy
* Patients who have received investigational drugs within 4 weeks prior to entry into this study or who have not recovered from side effects of such therapy
* Patients who are pregnant or breast feeding, or adults of reproductive potential not employing an effective method of birth control
* Concurrent severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, congestive cardiac failure, myocardial infarction within 6 months, poorly controlled hypertension, history of labile hypertension, history of poor compliance with antihypertensive regimen, chronic renal disease, or active uncontrolled infection) which could compromise participation in the study
* Acute or chronic liver disease (e.g., hepatitis, cirrhosis)
* Confirmed diagnosis of HIV infection
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of PTK787/ZK222584 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, bowel obstruction, or inability to swallow the capsules/tablets)
* Patients who are taking Coumadin (warfarin sodium); heparin is acceptable.
* Patients unwilling to, or unable to, comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-09; Primary Completion 2007-09 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Response rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Heikki Joensuu, M.D., Principal Investigator — Department of Oncology, Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland